CLINICAL TRIAL: NCT03180476
Title: Maintenance Therapy of Apatinib After Chemoradiotherapy in Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Mei Feng, Associate chief physician, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-NC-201701
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental): apatinib,500mg,qd，28 day/cycle until the emergence of PD, death, intolerable toxicity
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib, also known as YN968D1, is a tyrosine kinase inhibitor that selectively inhibits the vascular endothelial growth factor receptor-2 (VEGFR2, also known as KDR). It is an orally bioavailable, small molecule agent which is thought to inhibit angiogenesis in cancer cells; specifically apatinib inhibits VEGF-mediated endothelial cell migration and proliferation thus blocking new blood vessel formation in tumor tissue. This agent also mildly inhibits c-Kit and c-SRC tyrosine kinases.
  Other Names: YN968D1; apatinib mesylate tablets

SUMMARY:
The study is to evaluate the efficacy and safety of Apatinib as maintenace therapy for Nasopharyngeal Carcinoma With Metastasis after Chemoradiotherapy, including progress free survival(PFS)、overall survival (OS)、Quality of life score (QoL) and evaluation of drug safety.

DETAILED DESCRIPTION:
In locally advanced nasopharyngeal carcinoma(NPC), although radiotherapy and chemotherapy has been given, patients still locally recurrence and distant metastasis. There is no standard treatment recommendation for metastatic NPC who failed to chemoradiotherapy therapy. Apatinib has been approved as a second-line treatment for advanced gastric cancer. Several phase III studies of liver cancer, non small cell lung cancer and other tumors also showed apatinib has less toxicities and better tolerance. However, the clinical application of apatinib in nasopharyngeal carcinoma is still lack of evidence-based medicine. And this trial is designed to investigate the efficacy and safety of apatinib as maintenance therapy after chemoradiotherapy in nasopharyngeal carcinoma with metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ranging from 18 to 75 years old.
* Naive or recurrent Nasopharyngeal Carcinoma with metastasis after chemotherapy or radiotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* Adequate hematologic (neutrophil count>=1.5×109/L, hemoglobin>=80g/L, platelets>=80×109/L), hepatic function (aspartate transaminase (AST) & alanine transaminase(ALT) =<upper normal limit(UNL) x2, bilirubin level =< UNL x 1.5).
* Adequate renal function (creatinine clearance ≥ 60 mL/min).
* Patients have the ability to understand and voluntarily sign the informed consent, and allow adequate follow-up.

Exclusion Criteria:

* Previously, patients did receive the therapy of Apatinib or other VEGFR inhibitor, such as Sorafenib, Sunitinib.
* Difficulties in taking pills (inability to swallow tablets,GI tract resection, chronic bacillary diarrhea and intestinal obstruction).
* Bleeding tendency or coagulation disorders.
* with brain metastases.
* Uncontrolled hypertension (systolic pressure>150 mmHg , or diastolic pressure> 90 mmHg).
* Urine protein≥++, or urine protein in 24 hours≥1.0g
* Severe uncured wounds, ulcers or fracture.
* Pregnant or breast-feeding.
* Patients with epilepsy who need to take medicine (such as steroids or anti epilepsy agents).
* Patients have these symptoms, such as neurological diseases, mental illness, serious infection.
* The researcher believe that the Patient is not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  The first day of treatment to the date that disease progression is reported

SECONDARY OUTCOMES:
Overall survival | up to 24 months
  the first day of treatment to death or last survival confirm date.
Quality of Life (QoL) questionnaire | up to 24 months
  in cancer patients and survivors with dermatologic conditions. This is a nontherapeutic and nondiagnostic protocol to obtain quality of life assessments from cancer patients and survivors who have dermatologic conditions, whether related to cancer therapies, or directly related to the primary cancer diagnosis. Data will be collected by using one or more dermatology-specific QoL instruments based on the underlying skin condition/s.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Feng, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided